CLINICAL TRIAL: NCT02915146
Title: A Randomised Assessor-blinded Study to Compare Narrowband Ultraviolet B With Combined Narrowband Ultraviolet B and Ultraviolet A1 for Atopic Eczema
Brief Title: Narrowband Ultraviolet B Versus Narrowband Ultraviolet B Plus Ultraviolet A1 for Atopic Eczema
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Dundee (Other)
Collaborators: NHS Tayside (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2015DS04
Record Dates: First submitted 2016-08-04; First posted 2016-09-26 (Estimated); Last update posted 2020-11-06 (Actual); Status verified 2020-11

CONDITIONS: Atopic Eczema
Keywords: eczema; phototherapy; uva1; uvb; adults; children
MeSH Terms: conditions — Dermatitis, Atopic; Eczema

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- NB-UVB monotherapy (Active Comparator): Narrowband ultraviolet B monotherapy will be used
  Interventions: Radiation: combined ultraviolet phototherapy (NB-UVB + UVA1) vs. NB-UVB monotherapy
- NB-UVB + UVA1 (Active Comparator): Narrowband ultraviolet B combined with ultraviolet A1 phototherapy will be used
  Interventions: Radiation: combined ultraviolet phototherapy (NB-UVB + UVA1) vs. NB-UVB monotherapy

INTERVENTIONS:
Radiation: combined ultraviolet phototherapy (NB-UVB + UVA1) vs. NB-UVB monotherapy — NB-UVB combined with UVA1

SUMMARY:
Narrowband ultraviolet B phototherapy is the "standard" phototherapy for atopic eczema; ultraviolet A1 is sometimes used but is not a widely available treatment. We do not know the most important chromophores in treating atopic eczema; in which phototherapy is thought to work by improving epidermal barrier function, having beneficial effects on skin microbiome and local immunosuppression. It seems plausible that there are several chromophores and that 'targetting' several at once with different wavebands should help and for severe eczema that has not responded adequately to narrowband UVB or ultraviolet A1 alone the combination is sometimes used. This study is to test if the combination is moderately to greatly more effective than narrowband ultraviolet B monotherapy amongst patients referred for any form of first-line phototherapy for atopic eczema.

DETAILED DESCRIPTION:
Narrowband ultraviolet B phototherapy is the "standard" phototherapy widely used for atopic eczema; ultraviolet A1 is sometimes used but is not a widely available treatment. We do not know the most important chromophores in treating atopic eczema; in which phototherapy is thought to work by improving epidermal barrier function, having beneficial effects on skin microbiome and local immunosuppression.

It seems plausible that there are several chromophores (the molecules that absorb the ultraviolet photons to set in chain the effects we are aiming for) and that 'targetting' several chromophores at once with different wavebands should help. For severe eczema that has not responded adequately to narrowband UVB or ultraviolet A1 alone the combination is sometimes used in the few centres where UVA1 is available.

This study is to test if the combination is moderately to greatly more effective than narrowband ultraviolet B monotherapy amongst patients referred for any form of first-line phototherapy for atopic eczema.

ELIGIBILITY:
Inclusion Criteria:

* Patients with atopic eczema as diagnosed by a dermatologist, defined according to the UK Working Party diagnostic criteria, considered for any form of whole body phototherapy
* Age 12 years and above
* Able to understand and comply with protocol requirements and treatment visits, instructions and protocol stated restrictions
* Provision of written informed consent in accordance with the Scottish Children's Network consent guidance and standard operating procedure (SOP) for subjects aged 12-15 years
* Provision of written informed consent (subjects age 16 years and over)

Exclusion Criteria:

* Unable to provide written informed consent in accordance with the Scottish Children's Network consent guidance and SOP
* Unable to provide written informed consent (subjects age 16 years and over)
* Currently being treated, or treated within the past 2 weeks, with systemic immunosuppressive therapy
* Current use of drugs known to cause photosensitivity
* Phototherapy, photochemotherapy, or sunbed use in the preceding 3 months
* Known abnormal photosensitivity
* Previous history of skin cancer
* Participation in another research study within the past three months

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2020-08-26 (Actual); Study Completion 2020-08-26 (Actual)

PRIMARY OUTCOMES:
Change in EASI (eczema severity score) - proportions reaching 50% reduction | From beginning to end of treatment (25 weeks)
  observer-assessed eczema severity

SECONDARY OUTCOMES:
POEM (patient orientated eczema measure) | 26 weeks after treatment completion
  patient-assessed eczema severity

CONTACTS AND LOCATIONS:
Overall Officials: Robert S Dawe, Principal Investigator — NHS Tayside and University of Dundee
Locations (1):
- Ninewells Hospital, Dundee, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes